CLINICAL TRIAL: NCT02873650
Title: A Phase I, Open Label, Multicenter, Single Dose Study to Evaluate the Pharmacokinetics of Dabrafenib in Healthy Subjects With Normal Hepatic Function and Subjects With Impaired Hepatic Function
Brief Title: Pharmacokinetics of Dabrafenib in Subjects With Hepatic Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to continued enrolment difficulties.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CDRB436A2107
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-04

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; Healthy volunteers; Clinical pharmacology study; DRB436; dabrafenib; normal hepatic function; impaired hepatic function
MeSH Terms: interventions — dabrafenib

STUDY DESIGN:
Intervention Model Description: open-label, parallel group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 - Control group (Experimental)
  Interventions: Drug: dabrafenib
- Group 2-Moderate hepatic impairment (Experimental)
  Interventions: Drug: dabrafenib
- Group 3-Severe hepatic impairment (Experimental)
  Interventions: Drug: dabrafenib

INTERVENTIONS:
Drug: dabrafenib — Single dose of 100 mg dabrafenib on Day 1
  Other Names: DRB436

SUMMARY:
To characterize the pharmacokinetics and safety of dabrafenib following a single 100 mg oral dose in subjects with moderate and severe hepatic impairment.

ELIGIBILITY:
Inclusion criteria (for all subjects)

* Male and/or female subjects 18-75 years of age
* Females must be of non-childbearing potential . All non-postmenopausal females must have a confirmed negative serum pregnancy
* Subjects in good health condition as determined by no clinically significant findings from medical history and physical examination.
* Body mass index (BMI) between ≥18.0 and ≤38.0 kg/m2, with body weight ≥ 50 kg and no more than 140 kg
* Laboratory values must be within normal limits (correction allowed) or considered clinically insignificant
* Do not participate in any other clinical trials with a BRAF or other RAF inhibitors

Additional inclusion criteria for patients with normal hepatic function (Control group):

* Absence of clinically significant deviation from normal in medical history, physical examination, vital signs, electrocardiograms and clinical laboratory determinations.
* Must match to at least one hepatic impairment subject by age, gender and bodyweight

Additional inclusion criteria for hepatic impaired subjects:

* Confirmed hepatic disease
* Stable Child-Pugh status within 28 days prior to dosing.

Exclusion criteria for all subjects

* Participation in any clinical investigation within 4 weeks prior to dosing
* Significant acute illness within the two weeks prior to dosing
* History of immunodeficiency diseases, including a positive HIV
* History of malignancy of any organ system, treated or untreated, within 5 years
* Any prior history of keratoacanthoma and/or cutaneous squamous cell carcinoma
* A known diagnosis of any of the RASopathies, such as NF-1, Noonan syndrome, or related conditions.
* History of drug or alcohol abuse within the 6 months prior to dosing
* Smoking: urine cotinine levels below 500 ng/mL on Day -1.
* Use of drugs known to affect CYP3A4 and/or CYP2C8 including both (strong or moderate) inhibitors and inducers, within 7 days prior to dosing
* Administration of medications that prolong the QT interval within 4 weeks prior to dosing and until EOT.
* History or current diagnosis of cardiac disease indicating significant risk of safety
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs.

Additional exclusion criteria for healthy subjects (control group):

* Clinical evidence of liver disease or liver injury
* History or presence of renal impairment as indicated by abnormal creatinine or BUN values
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody

Additional exclusion criteria for subjects with hepatic impairment:

* Alcohol or drug abuse within one month prior to dosing or evidence of such
* History of liver transplantation at any time in the past and is on immunosuppressant therapy.
* Encephalopathy Grade 3 or worse within 28 days of dosing.
* History of surgical portosystemic shunt.
* Life expectancy ≤3 months

Other protocol-defined inclusion/exclusion may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Predose through 96 hours postdose
Area under the curve (AUClast) | Predose through 96 hours postdose
Area under the curve (AUFinf) | Predose through 96 hours postdose
Systemic drug clearance (CL/F) | Predose through 96 hours postdose
Time to reach maximum concentration (Tmax) | Predose through 96 hours postdose
Terminal elimination rate (Lambda_z) | Predose through 96 hours postdose
Elimination half-life (T1/2) | Predose through 96 hours postdose
Volume of distribution (Vz/F) | Predose through 96 hours postdose

SECONDARY OUTCOMES:
Number of subjects with adverse events | Time of study drug administration through 30 days postdose
Number of subjects with abnormal lab values related to study drug | Time of study drug administration through 30 days postdose
Number of subjects with abnormal blood pressure related to study drug | Time of study drug administration through 30 days postdose
Number of subjects with abnormal pulse rate related to study drug | Time of study drug administration through 30 days postdose
Number of subjects with abnormal respiratory rate related to study drug | Time of study drug administration through 30 days postdose
Number of subjects with abnormal body temperature related to study drug | Time of study drug administration through 30 days postdose
Changes in electrocardiogram (ECG) | Time of study drug administration through 30 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - American Institute of Research, Los Angeles, California
  - Omega Research Consultants LLC, DeBary, Florida
  - Hassman Research Institute, Berlin, New Jersey
  - Wake Research Associates Oncology, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17618